CLINICAL TRIAL: NCT03331120
Title: Addition of 3D Posture Corrective Orthosis To A Multimodal Program In The Treatment Of Nonspecific Neck Pain. A Randomized Pilot Trial.
Brief Title: Addition of 3D Posture Corrective Orthosis to A Multimodal Program of Treatment Of NSNP.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Samir Abdelkhalik Youssef, Principal Investigator, PHD Student at Department of Rehabilitation Medicine and Physical Therapy,Tongji Medical College,HUST,CHINA , Assistant Lecturer at Faculty of Physical Therapy - Beni-Suef University,Egypt., Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-2017
Record Dates: First submitted 2017-10-22; First posted 2017-11-06 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Neck Pain
Keywords: Neck pain; Ambulatory; Orthotic
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: A pilot double-blind randomized controlled trial, 24 patients will be randomized into two groups (study and control) using random number generator. The both groups will receive conventional treatment consisting of moist hot pack, soft tissue mobilization, manual therapy, therapeutic exercise. Additionally, the study group will receive ambulatory mirror image functional re-training through wearing 3D adjustable CTPCO.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): 1--Control group
  . Conventional treatment:
  1. moist hot pack.
  2. manual therapy.
  3. Therapeutic Exercise.
  4. Home program routine.
  Interventions: Device: ambulatory mirror image functional re-training through wearing 3D adjustable cervicothoracic Posture Corrective Orthotic(CTPCO)
- Study or Experimental Group (Experimental): 2--Experimental or study group:
  1. moist hot pack.
  2. manual therapy.
  3. Therapeutic Exercise.
  4. Home program routine.
  5. ambulatory mirror image functional re-training through wearing 3D adjustable cervical thoracic Posture Corrective orthosis (CTPCO) For 10 weeks(3Times/week for 20 minutes).
  Interventions: Device: ambulatory mirror image functional re-training through wearing 3D adjustable cervicothoracic Posture Corrective Orthotic(CTPCO)

INTERVENTIONS:
Device: ambulatory mirror image functional re-training through wearing 3D adjustable cervicothoracic Posture Corrective Orthotic(CTPCO) — Ambulatory a mirror image functional re-training This way of functional training will deliver via the use of adjustable cervicothoracic orthosis with the patient walking at approximately 2-3 miles per hour on a standard, motorized treadmill. The brace will reverse the abnormal posture according to the 3D posture analysis data. To facilitate tissue remodeling by reverse posture training, this called mirror image exercise.then the ambulatory exercises by using treadmill will be performed while the patient's mirror image posture will be held by the adjustable orthosis, ambulatory exercises for 20 minutes by using treadmill Based on Harrison et al and Hawes et al., approach, this program will be repeated 3 Times /week for 10 weeks.
  Other Names: moist hot pack; manual therapy; Therapeutic exercise; Home program routine

SUMMARY:
Nonspecific neck pain (NSNP) is one of the most common musculoskeletal problems treated by orthopaedic physicians and physiotherapists . NSNP has an annual incidence rate of 38 to 73% and a lifetime prevalence of approximately 48%, leading to both economic and social problems.

DETAILED DESCRIPTION:
Posture has emerged as a major risk factor associated with NSNP, but most previous studies have ignored correct posturing as an effective treatment. The few studies that used posture corrective strategies were based on a dated concept that did not incorporate the 3D nature of posture into the treatment strategy . Therefore, one of the major challenges faced by clinicians is how to incorporate 3D posture findings into the treatment plan.

Harrison and colleagues reported that posture problems occurred in the head, ribs and pelvis in three dimensions in the form of translations and rotational displacements. Therefore, we should consider three-dimensional postural assessment and correction during the treatment of NSNP to obtain long-lasting effects and prevent the recurrence of neck pain.

Several tools are available for objective postural measurements in clinical use, including simple plumb line measure, photographic techniques , moiré topography and various computer-assisted methods, such as electro goniometers. These methods are used in clinical assessments, but they have limitations, including the inability to measure neck posture as rotations and translations in six degrees of freedom, as mentioned by Harrison and colleagues.

The current study will use a 3D analysis system called the Global Postural System (GPS) , which is a novel device that investigates all postural variables at once and provides the managing physiotherapist with radiation-free and accurate measurements . This device also provides further information about foot pressure analysis and other 3D features that allow bracing designs to be tailored for each patient .

Numerous studies have shown that mirror images in motion exercises, which are prescribed specifically to help normalize the patient's neuromuscular dysfunction and postural deformation via reflecting the patient's posture across different planes, are more beneficial than a less personalized programme.

With these considerations in mind and to integrate the findings of 3D postural assessment into the treatment programme, we designed an adjustable cervico thoracic posture corrective orthotic (CTPCO) to be worn by the patient for a short time. The device has the ability to reflect all transitional displacements and rotational movements of the head. Ambulatory exercises will be performed using a treadmill while the CTPCO holds the patient's reverse posture.

We designed a randomized two-arm pilot trial to investigate the hypothesis that the addition of a 3D adjustable CTPCO to a multimodal programme will produce short- and long-term improvement effects on NSNP management outcomes (i.e., neck pain, neck disability and 3D posture parameters of the head).

The primary aim of this study is to evaluate the feasibility of conducting a larger randomized trial that considers recruitment, compliance to study protocols and adverse events. The secondary aim is to investigate the effect size of the addition of ambulatory mirror image functional re-training via the wearing of a 3D adjustable CTPCO compared to control group interventions for neck pain, disability and 3D posture parameters.

ELIGIBILITY:
Inclusion criteria

1. Male and female subjects age from 17 to 40 years
2. Neck pain with equal or greater than 3/10 on a visual analogue scale (VAS) and pain lasting more than 3 months (chronic neck pain) [26, 27]
3. Patients with neck disability; this is defined by a score of at least 5 (on a 50-point scale) on the neck disability index (NDI) [28]
4. Patients will be included if they have posture abnormalities by screening test using GPS at least 2 posture abnormalities.
5. Subjects must be able to continue treatment for 10 weeks and then attend 3-month follow-up
6. If patients can accept and sign informed consent form

Exclusion criteria

1. If patient report any of the following conditions:

   Neck pain associated with whiplash injuries, medical red flag history (such as tumour, fracture, metabolic diseases, rheumatoid arthritis and osteoporosis) [27].
2. Neck pain with cervical radiculopathy or neck pain associated with externalized cervical disc herniation [27]
3. Fibromyalgia syndrome; to avoid the similarity of fibromyalgia with a NSNP diagnosis, a physician will use the criteria for the clinical diagnosis of fibromyalgia according to the American College of Rheumatology [29]
4. If the patient had previous surgery in the neck area (irrespective of the reason for the operation) [27]
5. Neck pain accompanied by vertigo caused by vertebra basilar insufficiency or accompanied by non-cervicogenic headaches [27]
6. People will also be excluded if they are undergoing any type of pain treatment or they have psychiatric disorders or other problems that contraindicate the use of the techniques in this study [27]
7. If patient has true leg length discrepancy and an associated pathology of upper and lower limbs that may interfere with the global posture (e.g., foot, knee or hip deformities)
8. The patients will be unable to attend a 10-week treatment programme and follow-up assessments after 3 months

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
questionnaire to assess Feasibility. | Pre treatment at 1st day , post treatment after 10 weeks .
  Feasibility to assess feasibility of conducting future RCT.

SECONDARY OUTCOMES:
The Numeric Pain Rating Scale | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 3 months.
  is an 11-point numeric pain intensity ranging from 0 ('no pain') to 10 ('as much pain as possible'). A change of two points or more was identified as the minimal clinically an important difference in patients with chronic neck pain.
Neck Disability Index, Assess change of neck disability at baseline, after 10 weeks treatment and after 3 months follow up. | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 3 months.
  The NDI is a modification of the Oswestry Low Back Pain Disability Index. It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. The NDI has sufficient support and usefulness to retain its current status as the most commonly used self-report measure for neck pain The NDI can be scored as a raw score [2]or doubled and expressed as a percent [3]. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. All the points can be summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.
  0 points or 0% means no activity limitations, 50 points or 100% means complete activity limitation.
Three-dimensional posture parameters measured by GPS device. Assess change of posture parameters before, after treatment 10 weeks and after follow up 3 months. | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 3 months.
  Postural translation of head
  1. Tx(medio lateral translation )
  2. Tz(antero posterior translation )
  Postural rotations of head
  1. Rx(flexion or extension position)
  2. Ry (r.t rot. Or l.t rot.)
  3. RZ (r.t side bending or l.t side bending)
Active cervical ROM using CROM. | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 3 months.
  with an inclinometer (CROM Deluxe model, Performance Attainment Associates, Lindstrom, Minnesota).
  The CROM consists of 2 gravity-dependent goniometers, one compass dial, and a head-mounted frame allowing measurement of ROM in 3 planes (flexion/ extension, lateral flexion, rotation). A magnetic yoke consisting of 2 bar magnets held anteriorly and posteriorly was provided to reduce the influence of thoracic rotation. The CROM has demonstrated good concurrent validity for active ROM. According to the systematic review by Chen et al, the mean normative values of cervical ROM were determined to be: 52 degrees for flexion, 71 degrees for the extension, 72 degrees for rotation, and 43 degrees for lateral flexion. Documentation of cervical ROM was rendered in the form of the full range (ie, a total value for the sagittal, frontal, or transverse plane, yielding 3 measurements).
Zung Self-Rating Anxiety Scale (SAS) | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 3 months.
  The SAS test is self-administered, with each response using a 4-point scale, from 'none of the time" to "most of the time." There are 20 questions with 15 increasing anxiety level questions and 5 decreasing anxiety questions. There are two formats, self-evaluations and clinical evaluations.
Zung Self-Rating Depression Scale (SDS) | Pre treatment at 1st day , post treatment after 10 weeks , follow up after 3 months.
  scoring the SDS, a value of 1, 2, 3 and 4 is assigned to a response depending upon whether the item is worded positively or negatively. For items 1, 3, 4, 7, 8, 9, 10, 13, 15, 19 the scoring is:• A little of the time = 1• Some of the time = 2• Good part of the time = 3• Most of the time = 4 Items 2, 5, 6, 11, 12, 14, 16, 17, 18, 20 are reverse scored as follows:• Most of the time = 1• Good part of the time = 2• Some of the time = 3• A little of the time = 4 The SDS index is derived by dividing the sum of the values (raw scores) obtained on the 20 items by the maximum possible score of 80, and expressed as a decimal point.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Huang, Professor, Study Director — Tongji Hospital
Locations (1):
- Tongji Medical College, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
it is according to the opinion of my supervisor and also for the honesty of patients data as ethics it is not good to share its data in public. so we will see this issue at the end of study/

REFERENCES:
- [Derived] Youssef ASA, Xia N, Emara STE, Moustafa IM, Huang X. Addition of a new three-dimensional adjustable cervical thoracic orthosis to a multi-modal program in the treatment of nonspecific neck pain: study protocol for a randomised pilot trial. Trials. 2019 Apr 29;20(1):248. doi: 10.1186/s13063-019-3337-0. PMID 31036033
- Available data/document: Study Protocol: Neck pain,Ambulatory,Orthotic — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-019-3337-0 — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-019-3337-0